CLINICAL TRIAL: NCT00256451
Title: Defining an Endophenotype for Alcohol Misuse: A Focus On Minority Populations
Brief Title: Endophenotype for Alcohol Misuse in Healthy Minority Populations
Acronym: DEFINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, David Oslin, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 803866
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Naltrexone; Alcohol
MeSH Terms: interventions — Naltrexone; Ethanol; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ALC and NAL (Experimental): alcohol and active naltrexone
  Interventions: Drug: Naltrexone; Other: alcohol
- Sham ALC and NAL (Active Comparator): "sham" alcohol and active naltrexone
  Interventions: Drug: Naltrexone; Other: Sham alcohol
- placebo pill and ALC (Placebo Comparator): placebo naltrexone and alcohol
  Interventions: Drug: placebo; Other: alcohol
- placebo pill and Sham ALC (Placebo Comparator): placebo naltrexone and placebo (non-alcoholic) alcohol
  Interventions: Drug: placebo; Other: Sham alcohol

INTERVENTIONS:
Drug: Naltrexone — 50 mg/day for two days prior to the alcohol challenge session
  Other Names: ReVia
  Arms: ALC and NAL; Sham ALC and NAL
Drug: placebo — placebo pills
  Arms: placebo pill and ALC; placebo pill and Sham ALC
Other: alcohol — 190 proof alcohol prepared to 11% volume mixed with fruit juice.
  Arms: ALC and NAL; placebo pill and ALC
Other: Sham alcohol — non-alcoholic placebo alcohol
  Arms: Sham ALC and NAL; placebo pill and Sham ALC

SUMMARY:
The purpose of the study is to understand the relationship between what an individual inherited from their family (genetics), how they respond and feel after drinking alcohol, and how they respond to pre-treatment with naltrexone, a medication that blocks some of the effects of alcohol and is approved for the treatment of alcoholism. The investigators are conducting this study on those of African descent because there is almost no research focused on this group and the association with genetics. The investigators seek to enroll 40 people in the study. Participation will consist of 4 different alcohol challenge sessions in a cross over design. Each session will be separated by at least 10 days. In total, there will be four challenge sessions.

DETAILED DESCRIPTION:
We propose to test the degree to which specific genetic markers alter the relationship between subjective and objective measures of response to alcohol ingestion among non-alcohol dependent adults of African descent in a laboratory environment. To meet this aim, non-alcohol dependent adults of African descent will be recruited for participation to meet the N-goal of 40 trial completers. After consenting, genotyping, and completing the baseline assessment, they will participate in four separate alcohol challenge sessions separated by at least 10 days. During each of the sessions, subjects will be administered alcohol or sham drinking challenge sessions and pretreatment with either naltrexone (50 mg/day) or placebo in a double-blind fashion. The order of the four sessions will be randomly assigned. During each session, physiological and subjective response will be measured. We will select subjects to assure equal number of participants with at least one copy of the Val6 allele compared to those homozygous for the Ala6 allele.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and 21 years of age or older
* Drinks less than an average of 21 drinks/week with no more than 2 binge episodes per week
* Of African descent by self report

Exclusion Criteria:

* Meets DSM-IV criteria for lifetime dependence on any substance other than nicotine
* Subjects who test positive on the urine drug screen for opioids, cocaine, marijuana, or amphetamine at the screening visit
* Subjects who meet current or lifetime DSM-IV criteria for bipolar affective disorder, schizophrenia, or any psychotic disorder
* The presence of unstable or serious medical illness; including history of stroke, seizure disorder, severe liver disease (AST or ALT > 5X normal at the time of randomization), or unstable cardiac disease
* Needs treatment with any psychotropic medication (antidepressant, antipsychotic, benzodiazepine, or mood stabilizing medication)
* Pre-menopausal female subjects who are pregnant, nursing, or not using a reliable method of contraception
* Insulin-dependent diabetes
* Any medical or psychological condition that could jeopardize the subject's safe participation in the trial as determined by the PI.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Oslin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only randomized to 4 sequences and not to all 12 possible sequences.
Groups:
- Ntx-Alc; Placebo-Sham; Ntx-Sham; Placebo-Alc: Session1: alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
  Session2:placebo naltrexone and placebo (non-alcoholic) alcohol placebo: placebo pills Sham alcohol: non-alcoholic placebo alcohol Session3: "sham" alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session Sham alcohol: non-alcoholic placebo alcohol Session4: placebo naltrexone and alcohol placebo: placebo pills alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
- Ntx-Sham; Ntx-Alc; Placebo-Alc; Placebo-Sham: Session1: "sham" alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session Sham alcohol: non-alcoholic placebo alcohol Session2: alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
  Session3: placebo naltrexone and alcohol placebo: placebo pills alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
  Session4: placebo naltrexone and placebo (non-alcoholic) alcohol placebo: placebo pills Sham alcohol: non-alcoholic placebo alcohol
- Placebo-Alc; Ntx-Sham; Placebo-Sham; Ntx-Alc: Session1: placebo naltrexone and alcohol placebo: placebo pills alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
  Session2: "sham" alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session Sham alcohol: non-alcoholic placebo alcohol Session3:placebo naltrexone and placebo (non-alcoholic) alcohol placebo: placebo pills Sham alcohol: non-alcoholic placebo alcohol Session4: alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
- Placebo-Sham; Placebo-Alc; Ntx-Alc; Ntx-Sham: Session1: placebo naltrexone and placebo (non-alcoholic) alcohol placebo: placebo pills Sham alcohol: non-alcoholic placebo alcohol Session2: placebo naltrexone and alcohol placebo: placebo pills alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
  Session3: alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session alcohol: 190 proof alcohol prepared to 11% volume mixed with fruit juice.
  Session4: "sham" alcohol and active naltrexone Naltrexone: 50 mg/day for two days prior to the alcohol challenge session Sham alcohol: non-alcoholic placebo alcohol
Period: Session1
Arm/Group | Ntx-Alc; Placebo-Sham; Ntx-Sham; Placebo-Alc | Ntx-Sham; Ntx-Alc; Placebo-Alc; Placebo-Sham | Placebo-Alc; Ntx-Sham; Placebo-Sham; Ntx-Alc | Placebo-Sham; Placebo-Alc; Ntx-Alc; Ntx-Sham
Started (Crossover design: no of subjs who completed the PRIOR session) | 10 | 11 | 11 | 11
Completed | 10 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Session2
Arm/Group | Ntx-Alc; Placebo-Sham; Ntx-Sham; Placebo-Alc | Ntx-Sham; Ntx-Alc; Placebo-Alc; Placebo-Sham | Placebo-Alc; Ntx-Sham; Placebo-Sham; Ntx-Alc | Placebo-Sham; Placebo-Alc; Ntx-Alc; Ntx-Sham
Started (Crossover design: no of subjs who completed the PRIOR session) | 9 | 11 | 10 | 10
Completed | 9 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Session3
Arm/Group | Ntx-Alc; Placebo-Sham; Ntx-Sham; Placebo-Alc | Ntx-Sham; Ntx-Alc; Placebo-Alc; Placebo-Sham | Placebo-Alc; Ntx-Sham; Placebo-Sham; Ntx-Alc | Placebo-Sham; Placebo-Alc; Ntx-Alc; Ntx-Sham
Started (Crossover design: no of subjs who completed the PRIOR session) | 9 | 9 | 10 | 9
Completed | 9 | 9 | 10 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Session4
Arm/Group | Ntx-Alc; Placebo-Sham; Ntx-Sham; Placebo-Alc | Ntx-Sham; Ntx-Alc; Placebo-Alc; Placebo-Sham | Placebo-Alc; Ntx-Sham; Placebo-Sham; Ntx-Alc | Placebo-Sham; Placebo-Alc; Ntx-Alc; Ntx-Sham
Started (Crossover design: no of subjs who completed the PRIOR session) | 9 | 8 | 10 | 8
Completed | 9 | 8 | 10 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: all participants in the cross over study
Arm/Group | Overall Study Population
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 43
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Alcohol use [Mean (Standard Deviation); unit: total number of drinks in the week prior] — The average number of standard drinks per week prior to the trial.
  total number of drinks in the week prior | 3.2 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Biphasic Alcohol Effects Scale - Stimulation
Description: Change from baseline to peak for the feeling of stimulation after alcohol ingestion
  Biphasic Alcohol Effects Scale - Stimulation: sum of 7 items each rated on 11 point Likert scale (0=not at all, 10=extremely). Minimum=0, maximum=70, higher scores=worse outcome.
Time Frame: During challenge sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo ALC and NAL: "sham" alcohol and active naltrexone
  Naltrexone: 50 mg/day for two days prior to the alcohol challenge session
  Sham alcohol: non-alcoholic placebo alcohol
- Placebo Pill and Placebo ALC: placebo naltrexone and placebo (non-alcoholic) alcohol
  placebo: placebo pills
  Sham alcohol: non-alcoholic placebo alcohol
Arm/Group | ALC and NAL | Placebo ALC and NAL | Placebo Pill and ALC | Placebo Pill and Placebo ALC
Number analyzed (Participants) | 40 | 38 | 39 | 38
units on a scale | 11.3 (10.1) | 3.9 (5.1) | 8.7 (7.6) | 3.2 (4.6)

2. Primary Outcome: Profile of Mood States - Vigor
Description: Change from baseline to peak for the amount of Vigor experienced after alcohol ingestion
  Profile of Mood States - Vigor: sum of 6 items each rated on 5 point Likert scale (0: not at all, 4: extremely). Minimum=0, maximum=20, higher scores = better outcome
Time Frame: during the challenge session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALC and NAL | Placebo ALC and NAL | Placebo Pill and ALC | Placebo Pill and Placebo ALC
Number analyzed (Participants) | 40 | 38 | 39 | 38
units on a scale | 2.1 (2.5) | 1.1 (1.2) | 1.8 (1.4) | 1.2 (1.3)

3. Primary Outcome: Subjective High From Alcohol Scale
Description: Change from baseline to peak for the self reported feeling of being high after drinking
  Subjective High from Alcohol Scale: sum of 15 items rated on a 8 point Likert scale (0-7). Minimum=0, maximum=105, higher scores=worse outcomes
Time Frame: during the alcohol ingestion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALC and NAL | Placebo ALC and NAL | Placebo Pill and ALC | Placebo Pill and Placebo ALC
Number analyzed (Participants) | 40 | 38 | 39 | 38
units on a scale | 17.9 (17.2) | 4.5 (5.4) | 14.7 (13.1) | 2.7 (5.3)

4. Secondary Outcome: Biphasic Alcohol Effects Scale - Sedation
Description: Change from baseline to peak of the amount of sedation post ingestion of alcohol
  Biphasic alcohol effects scale - Sedation: sum of 7 items rated on 11 point Likert scale (0=not at all, 10=extremely). Minimum=0, maximum=70, lower scores=worse outcomes
Time Frame: During the challenge session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALC and NAL | Placebo ALC and NAL | Placebo Pill and ALC | Placebo Pill and Placebo ALC
Number analyzed (Participants) | 40 | 38 | 39 | 38
units on a scale | 14.8 (13.7) | 13.4 (16.1) | 15.9 (15.8) | 15.4 (16.3)

5. Secondary Outcome: Profile of Mood States - Fatigue Scale
Description: Change from baseline to peak of the degree of fatigue experienced after alcohol ingestion
  Profile of Mood States - Fatigue scale: sum of 5 items rated on 5-point Likert scale (0=not at all, 4=extremely). Minimum=0, maximum=20, higher score=worse outcome
Time Frame: During the challenge session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALC and NAL | Placebo ALC and NAL | Placebo Pill and ALC | Placebo Pill and Placebo ALC
Number analyzed (Participants) | 40 | 38 | 39 | 38
units on a scale | 2.2 (2.1) | 1.6 (1.4) | 2.0 (1.6) | 1.5 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during each session which typically occurred over 3 hours.
Description: We assessed for any adverse event reported related to the medication taken prior to the session or the alcohol during the session.
Arm/Group | ALC and NAL | Placebo ALC and NAL | Placebo Pill and ALC | Placebo Pill and Placebo ALC
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38 | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/39 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No